CLINICAL TRIAL: NCT02142998
Title: A Prospective Blinded Randomized Study Comparing Laparoscopic Sleeve Gastrectomy and Laparoscopic Roux-en-y Gastric Bypass and Their Effect on Gastro-Esophageal Reflux Disease Using 24 Horus pH Monitoring
Acronym: GERD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: On hold due to poor enrollment and high drop-out rate.
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mehran Anvari, Doctor, McMaster University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-001
Record Dates: First submitted 2014-03-24; First posted 2014-05-20 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: GERD
Keywords: GERD; Laparoscopic; sleeve; gastrectomy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GERD Symptoms (Active Comparator)
  Interventions: Other: 24 pH monitoring; Other: Esophageal Manometry:
- No GERD Symptoms (Active Comparator)
  Interventions: Other: 24 pH monitoring; Other: Esophageal Manometry:

INTERVENTIONS:
Other: 24 pH monitoring — The study is performed with the patient fasting for a minimum of 6 hours. A single channel or dual channel (15 cm spacing) pH probe is inserted trans nasally. The pH sensor, or distal pH sensor in the case of 2 channel testing, is positioned 5 cm above the proximal margin of the LES, as determined by esophageal manometric testing. pH-Z ambulatory monitor (Given Imaging Digitrapper) is used for data acquisition and the data analyzed with pH Analysis Program (Given Imaging AccuView). The number of reflux events, defined as a drop in esophageal pH readings below 4.0, is recorded and the percentage of time with esophageal acid exposure is analyzed using defined protocols and accepted normal values.
Other: Esophageal Manometry: — A high resolution esophageal manometry catheter is used for testing and inserted Trans nasally. The patient is given 10 liquid swallows (5mL of water), at intervals of approximately 30 seconds. The catheter (Sierra Scientific/Given Imaging) has 36 sensors, each one averaging pressures from 12 circumferential positions. This gives a total of 432 data points. The sensors are placed 1 cm apart, spanning a length of 35 cm. The catheter simultaneously records pressure readings from the esophagus, sphincter regions (UES and LES), pharynx and stomach without the need for a station pull-through technique. Results are reported according to defined protocols and accepted normal values.

SUMMARY:
Obesity has become a significant health problem in Canada. It is known to be a risk factor for many diseases, including Gastro-Esophageal Reflux Disease (GERD). When medical efforts to lose weight fail, patients often consider bariatric surgical procedures as the next step. The two most common bariatric procedures performed are Roux-en-Y Gastric Bypass (LRYGB) and Laparoscopic Sleeve Gastrectomy (LSG). The gold standard for diagnosing GERD is Esophageal pH monitoring, as it is the most objective method to document the reflux, assess the severity and monitor the response to treatment of the disease. In the last few years LSG has gained in popularity due to its simplicity and short operative time. Currently the comparison between bariatric surgery and GERD symptoms is very one sided. There are significant numbers of studies with conclusive results that state that LRYGB has a positive effect on GERD symptoms, however there is little evidence that states the same about LSG. This means that the relationship between LSG and GERD is inconclusive. An objective evaluation of GERD using 24 hour pH monitoring and validated CRFs at different follow up time points will contribute greatly to our understanding of what this relationship might be.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled criteria for bariatric surgery as coined by National Institutes of Health conference.
* Their age is ≥18 years and ≤70 years
* The group with symptoms of GERD needs to have diagnosis of GERD in their medical record and taking proton pump inhibitors on a daily basis.
* Able and willing to give written consent
* The patient is willing to perform the pre-operative tests required for this study.
* The patient fits for both surgeries - LSG or LRYGB

Exclusion Criteria:

* Previous bariatric surgery
* Previous anti reflux procedure
* Contra-indication to general anesthesia
* Any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Pregnant or lactating female (Women of child bearing potential must take a pregnancy test prior to surgery)
* Hiatal hernia above 4cm (measured in the pre-operative gastroscopy).
* Multiple surgeries in abdominal cavity or previous small bowel disease/resection
* Patient on CPAP treatment for his OSA disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Observe acid exposure to the distal esophagus | 1 year
  This will be measured using the esophageal 24 hours monitoring before surgery and at the 6 month follow up. The patients will be randomized to two different types of surgery and the results compared.

SECONDARY OUTCOMES:
Compare GERD symptoms in patients. | 1 year
  This will be measured using esophageal manometry prior to surgery and at the six month follow up visit. We are looking for time in minutes with a pH of below 4 and a Demeeser score of below 14.7

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Anvari, MB BS, PhD, Principal Investigator — Centre for Minimal Access Surgery, McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada